CLINICAL TRIAL: NCT01890759
Title: Immunogenicity and Safety of a Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) in Subjects Aged 9 to 23 Months in India and in the Russian Federation
Brief Title: Immunogenicity and Safety of Menactra® Vaccine in Subjects Aged 9 to 23 Months in India and in the Russian Federation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MTA70; U1111-1122-2171 (Other: WHO); CTRI/2014/12/005272 (Registry Identifier: Clinical Trials Registry - India)
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal Infection; Menactra®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Meningococcal Diphtheria Toxoid Vaccine (Experimental): Participants at age 9 to 17 months of enrollment will receive 2 doses on Menactra vaccine at 3 to 6 months apart
  Interventions: Biological: Meningococcal Diphtheria Toxoid Vaccine

INTERVENTIONS:
Biological: Meningococcal Diphtheria Toxoid Vaccine — 0.5 mL, Intramuscular
  Other Names: Menactra®

SUMMARY:
The purpose of this study is to assess the immunogenicity and safety of Menactra® vaccine given as a two-dose series in infants and toddlers.

Primary Objectives:

* To assess the seroprotection rate (percentage of subjects with a serum bactericidal assay using human complement [SBA-HC] titer ≥ 1:8) 28 days after the second of 2 doses of Menactra® administered 3 to 6 months apart.

Secondary Objectives:

* To assess the immune responses to meningococcal antigens (serogroups A, C, Y, and W-135) 28 days following the second vaccination with Menactra® using SBA-HC and SBA-BR titers.
* To assess the safety profile of Menactra® after each and any vaccination.

DETAILED DESCRIPTION:
Study participants will receive 2 doses on Menactra® vaccine at 3 to 6 months apart and will be monitored for safety and immunogenicity.

The planned duration of each subject's participation in the trial will be from 118 to 215 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 9 to 17 months on the day of inclusion
* Informed consent form has been signed and dated by the parent(s) or other legally acceptable representative(s) (if applicable)
* Subject and parent/legally acceptable representative (if applicable) able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in the 4 weeks preceding inclusion or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding each trial vaccination or planned receipt of any vaccine in the 4 weeks following each trial vaccination, except for:
* (i) influenza vaccination, which may be received at least 2 weeks before study vaccines.
* (ii) measles (M) or measles, mumps, rubella (MMR) routine vaccination, which can be administered concomitantly with the first dose of study vaccine as per routine immunization schedule
* (iii) for subjects enrolled at Indian sites: oral poliomyelitis vaccine (OPV) received during National Immunization Days (NIDs) and supplementary immunization activity days (SIADs)
* Previous vaccination against meningococcal disease with either the study vaccine or another meningococcal vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* History of meningococcal diseases, confirmed either clinically, serologically, or microbiologically
* At high risk, in the opinion of the Investigator, for meningococcal disease during the trial
* Known or suspected systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Known thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* In an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* For subjects enrolled at Indian sites: Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C).
* For subjects enrolled at Russian sites: Acute disease of any severity on the day of vaccination or febrile illness (axillary temperature ≥ 37.0°C).

A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.

* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* Personal history of Guillain-Barré Syndrome.

Ages: 9 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-06-25 (Actual); Primary Completion 2016-04-12 (Actual); Study Completion 2016-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (8):
- India (4):
  - Vadodara, Gujarat
  - Kolkata, West Bengal
  - Lucknow
  - Vellore
- Russia (4):
  - Murmansk
  - Perm
  - Saint Petersburg
  - Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 25 June 2013 to 05 November 2013 (Russian Federation) and 24 March 2015 to 17 November 2015 (India) at 4 clinic sites in Russia and 4 clinic sites in India.
Pre-assignment Details: A total of 300 participants (100 in Russia and 200 in India) were enrolled. Of the 100 Russians, 2 did not receive the second vaccination. Of the 200 Indians, 1 did not receive the first vaccination and 8 did not receive the second vaccination.
Groups:
- Russian Federation: Participants in the Russian Federation who received 1 dose of Menactra vaccine on Day 0 when 9 to 17 months of age and a second dose of Menactra vaccine no less than 3 months and no more than 6 months after the first injection.
- India: Participants in India who received 1 dose of Menactra vaccine on Day 0 when 9 to 17 months of age and a second dose of Menactra vaccine no less than 3 months and no more than 6 months after the first injection.
Period: Overall Study
Arm/Group | Russian Federation | India
Started | 100 | 200
Completed | 98 | 188
Not Completed | 2 | 12
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Russian Federation | India | Total
Number analyzed (Participants) | 100 | 200 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 200 | 300
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months]
  Age Continuous | 13.5 (2.7) | 12.9 (3.0) | 13.1 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 69 | 128
  Male | 41 | 131 | 172
Region of Enrollment [Number; unit: Participants]
  Russia | 100 | 0 | 100
  India | 0 | 200 | 200

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Seroprotection Using a Serum Bactericidal Assay Human Complement With Antibody Titers ≥ 1:8 for Meningococcal Serogroups A, C, Y, and W-135 Before and Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-HC assay. Seroprotection was defined as antibody titers ≥ 1:8.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-second vaccination
Population: Seroprotection was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A; Pre vaccination 1 (N=77,169) | 45.5 | 55.0
  Serogroup A; Post vaccination 2 (N=77,166) | 98.7 | 97.6
  Serogroup C; Pre vaccination 1 (N=77,169) | 6.5 | 4.7
  Serogroup C; Post vaccination 2 (N=77,169) | 92.2 | 95.9
  Serogroup Y; Pre vaccination 1 (N=77,169) | 5.2 | 6.5
  Serogroup Y; Post vaccination 2 (N=77,169) | 96.1 | 98.2
  Serogroup W 135; Pre vaccination 1 (N=77,169) | 7.8 | 5.3
  Serogroup W 135; Post vaccination 2 (N=77,169) | 100.0 | 99.4

2. Secondary Outcome: Percentage of Participants Achieving the Threshold Using a Serum Bactericidal Assay Human Complement With Antibody Titers ≥ 1:4 for Meningococcal Serogroups A, C, Y, and W-135 Before and Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-HC assay. The threshold was defined as antibody titers ≥ 1:4.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: The threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A; Pre vaccination 1 (N=77,169) | 88.3 | 97.6
  Serogroup A; Post vaccination 2 (N=77,166) | 100.0 | 99.4
  Serogroup C; Pre vaccination 1 (N=77,169) | 19.5 | 14.2
  Serogroup C; Post vaccination 2 (N=77,169) | 98.7 | 98.8
  Serogroup Y; Pre vaccination 1 (N=77,169) | 9.1 | 11.8
  Serogroup Y; Post vaccination 2 (N=77,169) | 98.7 | 100.0
  Serogroup W 135; Pre vaccination 1 (N=77,169) | 14.3 | 10.7
  Serogroup W 135; Post vaccination 2 (N=77,169) | 100.0 | 100.0

3. Secondary Outcome: Percentage of Participants With At Least Four-Fold Rise in Threshold in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers by Serum Bactericidal Assay Using Human Complement Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-HC assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: The threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A (N=77,166) | 90.9 | 84.9
  Serogroup C (N=77,169) | 76.6 | 92.3
  Serogroup Y (N=77,169) | 90.9 | 92.3
  Serogroup W 135 (N=77,169) | 90.9 | 97.0

4. Secondary Outcome: Percentage of Participants Achieving the Threshold in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers ≥ 1:8 by Serum Bactericidal Assay Using Human Complement Before and Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-HC assay. The threshold was defined as antibody titers ≥ 1:8.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: The threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A; Pre vaccination 1 (N=77,169) | 45.5 | 55.0
  Serogroup A; Post vaccination 2 (N=77,166) | 98.7 | 97.6
  Serogroup C; Pre vaccination 1 (N=77,169) | 6.5 | 4.7
  Serogroup C; Post vaccination 2 (N=77,169) | 92.2 | 95.9
  Serogroup Y; Pre vaccination 1 (N=77,169) | 5.2 | 6.5
  Serogroup Y; Post vaccination 2 (N=77,169) | 96.1 | 98.2
  Serogroup W-135; Pre vaccination 1 (N=77,169) | 7.8 | 5.3
  Serogroup W-135; Post vaccination 2 (N=77,169) | 100.0 | 99.4

5. Secondary Outcome: Percentage of Participants Achieving the Threshold in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers ≥ 1:8 by Serum Bactericidal Assay Using Baby Rabbit Complement Before and Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-BR assay. The threshold was defined as antibody titers ≥ 1:8.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A; Pre vaccination 1 (N=75,165) | 25.3 | 4.8
  Serogroup A; Post vaccination 2 (N=77,161) | 100.0 | 98.8
  Serogroup C; Pre vaccination 1 (N=76,166) | 5.3 | 10.8
  Serogroup C; Post vaccination 2 (N=77,166) | 97.4 | 94.0
  Serogroup Y; Pre vaccination 1 (N=76,166) | 84.2 | 84.3
  Serogroup Y; Post vaccination 2 (N=77,164) | 100.0 | 100.0
  Serogroup W-135; Pre vaccination 1 (N=76,165) | 27.6 | 18.2
  Serogroup W-135; Post vaccination 2 (N=77,163) | 100.0 | 100.0

6. Secondary Outcome: Percentage of Participants Achieving the Threshold in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers ≥ 1:4 by Serum Bactericidal Assay Using Human Complement Before and Following Vaccination With Menactra®
Description: as for outcome 2
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: The threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A; Pre vaccination 1 (N=77,169) | 88.3 | 97.6
  Serogroup A; Post vaccination 2 (N=77,166) | 100.0 | 99.4
  Serogroup C; Pre vaccination 1 (N=77,169) | 19.5 | 14.2
  Serogroup C; Post vaccination 2 (N=77,169) | 98.7 | 98.8
  Serogroup Y; Pre vaccination 1 (N=77,169) | 9.1 | 11.8
  Serogroup Y; Post vaccination 2 (N=77,169) | 98.7 | 100.0
  Serogroup W-135; Pre vaccination 1 (N=77,169) | 14.3 | 10.7
  Serogroup W-135; Post vaccination 2 (N=77,169) | 100.0 | 100.0

7. Secondary Outcome: Percentage of Participants Achieving the Threshold in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers ≥ 1:4 by Serum Bactericidal Assay Using Baby Rabbit Complement Before and Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-BR assay. The threshold was defined as antibody titers ≥ 1:4.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: The threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A; Pre vaccination 1 (N=75,165) | 26.7 | 5.5
  Serogroup A; Post vaccination 2 (N=77,161) | 100.0 | 98.8
  Serogroup C; Pre vaccination 1 (N=76,166) | 5.3 | 11.4
  Serogroup C; Post vaccination 2 (N=77,166) | 97.4 | 94.0
  Serogroup Y; Pre vaccination 1 (N=76,166) | 84.2 | 84.3
  Serogroup Y; Post vaccination 2 (N=77,164) | 100.0 | 100.0
  Serogroup W-135; Pre vaccination 1 (N=76,165) | 27.6 | 19.4
  Serogroup W-135; Post vaccination 2 (N=77,163) | 100.0 | 100.0

8. Secondary Outcome: Percentage of Participants With At Least Four-Fold Rise in Threshold Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers by Serum Bactericidal Assay Using Human Complement Following Vaccination With Menactra®
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: The threshold was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A (N=77,166) | 90.9 | 84.9
  Serogroup C (N=77,169) | 76.6 | 92.3
  Serogroup Y (N=77,169) | 90.9 | 92.3
  Serogroup W 135 (N=77,169) | 90.9 | 97.0

9. Secondary Outcome: Percentage of Participants With At Least Four-Fold Rise in Meningococcal Serogroups A, C, Y, and W-135 Antibody Titers by Serum Bactericidal Assay Using Baby Rabbit Complement Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-BR assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Percentage of participants
  Serogroup A (N=75,158) | 96.0 | 96.8
  Serogroup C (N=76,163) | 94.7 | 92.0
  Serogroup Y (N=76,161) | 68.4 | 66.5
  Serogroup W 135 (N=76,159) | 96.1 | 96.2

10. Secondary Outcome: Serum Bactericidal Assay Using Human Complement Antibody Geometric Mean Titers of Meningococcal Serogroups A, C, Y, and W-135 Before and Following Vaccination With Menactra®
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Titers (1/dil)
  Serogroup A; Pre vaccination 1 (N=77,169) | 5.73 [4.92 to 6.68] | 6.82 [5.94 to 7.83]
  Serogroup A; Post vaccination 2 (N=77,166) | 171 [126 to 232] | 95.2 [77.4 to 117]
  Serogroup C; Pre vaccination 1 (N=77,169) | 2.46 [2.20 to 2.75] | 2.50 [2.18 to 2.86]
  Serogroup C; Post vaccination 2 (N=77,169) | 49.3 [33.8 to 71.8] | 128 [102 to 160]
  Serogroup Y; Pre vaccination 1 (N=77,169) | 2.35 [2.04 to 2.72] | 2.49 [2.16 to 2.86]
  Serogroup Y; Post vaccination 2 (N=77,169) | 54.9 [41.3 to 73.0] | 104 [84.8 to 128]
  Serogroup W 135; Pre vaccination 1 (N=77,169) | 2.57 [2.15 to 3.08] | 2.45 [2.12 to 2.82]
  Serogroup W 135; Post vaccination 2 (N=77,169) | 114 [92.3 to 140] | 201 [167 to 241]

11. Secondary Outcome: Serum Bactericidal Assay Using Baby Rabbit Complement Geometric Mean Titers of Meningococcal Serogroups A, C, Y, and W-135 Before and Following Vaccination With Menactra®
Description: Functional antibody activity against the meningococcal serogroups A, C, Y, and W-135 antigens contained in Menactra vaccine was measured using a SBA-BR.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Titers (1/dil)
  Serogroup A; Pre vaccination 1 (N=75,165) | 6.47 [3.93 to 10.6] | 2.55 [2.16 to 3.02]
  Serogroup A; Post vaccination 2 (N=77,161) | 1940 [1612 to 2336] | 1426 [1165 to 1746]
  Serogroup C; Pre vaccination 1 (N=76,166) | 2.38 [2.00 to 2.82] | 3.27 [2.62 to 4.09]
  Serogroup C; Post vaccination 2 (N=77,166) | 326 [240 to 444] | 781 [577 to 1057]
  Serogroup Y; Pre vaccination 1 (N=76,166) | 87.3 [55.5 to 137] | 95.2 [71.7 to 126]
  Serogroup Y; Post vaccination 2 (N=77,164) | 734 [618 to 872] | 805 [669 to 968]
  Serogroup W 135; Pre vaccination 1 (N=76,165) | 5.66 [3.77 to 8.49] | 4.44 [3.40 to 5.80]
  Serogroup W 135; Post vaccination 2 (N=77,163) | 1260 [967 to 1640] | 1134 [913 to 1409]

12. Secondary Outcome: Serum Bactericidal Assay Using Human Complement Antibody Geometric Mean Titer Ratios of Meningococcal Serogroups A, C, Y, and W-135 Following Vaccination With Menactra®
Description: as for outcome 3
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titer ratios were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratios
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Titer ratios
  Serogroup A (N=77,166) | 29.8 [21.4 to 41.5] | 13.9 [10.8 to 18.1]
  Serogroup C (N=77,169) | 20.0 [13.8 to 29.2] | 51.3 [39.4 to 66.8]
  Serogroup Y (N=77,169) | 23.4 [16.6 to 32.8] | 41.9 [32.8 to 53.6]
  Serogroup W 135 (N=77,169) | 44.2 [32.7 to 59.8] | 82.2 [65.4 to 103]

13. Secondary Outcome: Serum Bactericidal Assay Using Baby Rabbit Complement Geometric Mean Titer Ratios of Meningococcal Serogroups A, C, Y, and W-135 Before and Following Vaccination With Menactra®
Description: as for outcome 9
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titer ratios were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer ratios
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 77 | 169
Titer ratios
  Serogroup A (N=75,158) | 305 [182 to 512] | 540 [416 to 700]
  Serogroup C (N=76,163) | 140 [97.4 to 202] | 240 [168 to 344]
  Serogroup Y (N=76,161) | 8.45 [5.50 to 13.0] | 8.50 [6.01 to 12.0]
  Serogroup W 135 (N=76,159) | 223 [137 to 365] | 246 [177 to 342]

14. Secondary Outcome: Percentage of Participants Reporting Solicited Injection Site or Systemic Reactions Following Each Vaccination With Menactra®
Description: Injection site: Tenderness, Erythema, and Swelling. Systemic: Fever (Temperature), Vomiting, Crying abnormal, Drowsiness, Appetite lost, Irritability. Grade 3 Injection site: Tenderness, Cries when injected limb is moved or the movement of the injected limb is reduced. Erythema and Swelling, ≥50 mm. Grade 3 Systemic: Fever, >39.5C; Vomiting, ≥6 episodes per 24 hours or requiring parenteral hydration; Crying abnormal, >3 hours; Drowsiness, Sleeping most of the time or difficult to wake; Appetite lost, Refuses ≥3 feeds/meals or refuses most feeds/meals; Irritability, Inconsolable.
Time Frame: Day 0 up to Day 7 post-each vaccination
Population: Solicited injection site and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Russian Federation | India
Number analyzed (Participants) | 100 | 199
Percentage of participants
  Any Inj. site Tenderness; Post dose 1; N=100,199 | 13.0 | 14.6
  Grade 3 Inj. site Tenderness;Post dose 1;N=100,199 | 0 | 0.5
  Any Inj. site Erythema; Post dose 1; N=100,199 | 28.0 | 4.5
  Grade 3 Inj. site Erythema; Post dose 1; N=100,199 | 1.0 | 0.5
  Any Inj. site Swelling; Post dose 1; N=100,199 | 8.0 | 3.5
  Grade 3 Inj. site Swelling; Post dose 1; N=100,199 | 0 | 0.5
  Any Inj. site Tenderness; Post dose 2; N=98,188 | 13.3 | 10.1
  Grade 3 Inj. site Tenderness;Post dose 2;N=98,188 | 0 | 0
  Any Inj. site Erythema; Post dose 2; N=98,188 | 16.3 | 2.1
  Grade 3 Inj. site Erythema; Post dose 2; N=98,188 | 2.0 | 0
  Any Inj. site Swelling; Post dose 2; N=98,188 | 7.1 | 2.7
  Grade 3 Inj. site Swelling; Post dose 2; N=98,188 | 1.0 | 0
  Any Fever; Post dose 1; N=100,197 | 0 | 7.1
  Grade 3 Fever; Post dose 1; N=100,197 | 0 | 0.5
  Any Vomiting; Post dose 1; N=100,199 | 2.0 | 9.5
  Grade 3 Vomiting; Post dose 1; N=100,199 | 0 | 0
  Any Crying abnormal; Post dose 1; N=100,199 | 8.0 | 12.6
  Grade 3 Crying abnormal; Post dose 1; N=100,199 | 0 | 0
  Any Drowsiness; Post dose 1; N=100,199 | 14.0 | 9.5
  Grade 3 Drowsiness; Post dose 1; N=100,199 | 0 | 0
  Any Appetite lost; Post dose 1; N=100,199 | 14.0 | 17.1
  Grade 3 Appetite lost; Post dose 1; N=100,199 | 0 | 1.5
  Any Irritability; Post dose 1; N=100,199 | 23.0 | 14.6
  Grade 3 Irritability; Post dose 1; N=100,199 | 0 | 0.5
  Any Fever; Post dose 2; N=98,185 | 6.1 | 7.0
  Grade 3 Fever; Post dose 2; N=98,185 | 0 | 0.5
  Any Vomiting; Post dose 2; N=98,188 | 0 | 7.4
  Grade 3 Vomiting; Post dose 2; N=98,188 | 0 | 0
  Any Crying abnormal; Post dose 2; N=98,188 | 9.2 | 9.6
  Grade 3 Crying abnormal; Post dose 2; N=98,188 | 0 | 0
  Any Drowsiness; Post dose 2; N=98,188 | 11.2 | 3.7
  Grade 3 Drowsiness; Post dose 2; N=98,188 | 1.0 | 0
  Any Appetite lost; Post dose 2; N=98,188 | 11.2 | 9.6
  Grade 3 Appetite lost; Post dose 2; N=98,188 | 1.0 | 0.5
  Any Irritability; Post dose 2; N=98,188 | 12.2 | 9.0
  Grade 3 Irritability; Post dose 2; N=98,188 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 up to Day 28 post-each vaccination and SAEs were collected throughout the study.
Arm/Group | Russian Federation | India
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/199
Serious Adverse Events (participants affected / at risk) | 1/100 | 3/199
Other Adverse Events (participants affected / at risk) | 35/100 | 40/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Russian Federation (N=100) | India (N=199)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Russian Federation (N=100) | India (N=199)
Injection site Tenderness (General disorders) | 24 (24) | 40 (40)
Injection site Erythema (General disorders) | 35 (35) | 12 (12)
Injection site Swelling (General disorders) | 13 (13) | 10 (10)
Fever (General disorders) | 6 (6) | 25 (25)
Crying abnormal (Psychiatric disorders) | 15 (15) | 33 (33)
Drowsiness (Nervous system disorders) | 22 (22) | 24 (24)
Appetite lost (Metabolism and nutrition disorders) | 21 (21) | 40 (40)
Irritability (Psychiatric disorders) | 29 (29) | 34 (34)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 10 (11)
Vomiting (Gastrointestinal disorders) | 2 (2) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications